CLINICAL TRIAL: NCT06251050
Title: A Lithium-containing Mouthwash Prevention and Treatment of Oral Mucositis and Dysgeusia in Patients Undergoing Radiotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-863
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Malignant Head and Neck Tumors
Keywords: head and neck squamous cell carcinoma; nasopharyngeal carcinoma; Malignant Head and Neck tumors; oral mucositis; lithium-containing mouthwash
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Nasopharyngeal Carcinoma; Stomatitis

STUDY DESIGN:
Intervention Model Description: Phase 1 containes 5 arms including 0.03, 0.06, 0.10, 0.15 and 0.30 mol/L lithium mouthwash.
  Phase 2 containes 2 arms including lithium mouthwash group and palcebo group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- 0.03 mol/L lithium mouthwash (Experimental): The main ingredients of mouthwash are lithium carbonate and citric acid, transparent colorless liquid. In this group, 10 ml of 0.03 mol/L lithium mouthwash is used to gargle and left in the mouth for 5 min to be spat out from the first day of radiotherapy up to the end of treatment.
- 0.06 mol/L lithium mouthwash (Experimental): The main ingredients of mouthwash are lithium carbonate and citric acid, transparent colorless liquid.. In this group, 10 ml of 0.06 mol/L lithium mouthwash is used to gargle and left in the mouth for 5 min to be spat out from the first day of radiotherapy up to the end of treatment.
- 0.10 mol/L lithium mouthwash (Experimental): The main ingredients of mouthwash are lithium carbonate and citric acid,transparent colorless liquid. In this group, 10 ml of 0.10 mol/L lithium mouthwash is used to gargle and left in the mouth for 5 min to be spat out from the first day of radiotherapy up to the end of treatment.
- 0.15 mol/L lithium mouthwash (Experimental): The main ingredients of mouthwash are lithium carbonate and citric acid, transparent colorless liquid. In this group, 10 ml of 0.15 mol/L lithium mouthwash is used to gargle and left in the mouth for 5 min to be spat out from the first day of radiotherapy up to the end of treatment.
- 0.30 mol/L lithium mouthwash (Experimental): The main ingredients of mouthwash are lithium carbonate and citric acid, transparent colorless liquid. In this group, 10 ml of 0.30 mol/L lithium mouthwash is used to gargle and left in the mouth for 5 min to be spat out from the first day of radiotherapy up to the end of treatment.
  Interventions: Drug: lithium-containing mouthwash
- Lithium mouthwash (Active Comparator): Effective lithium salt concentrations screened in the Phase I trial is used as active interventions in this group of interventions.
  Interventions: Drug: lithium-containing mouthwash
- Placebo mouthwash (Placebo Comparator): Placebo Mouthwash is mainly composed of citric acid and sodium hydroxide, transparent colorless liquid.
  Interventions: Drug: Plcacebo mouthwash

INTERVENTIONS:
Drug: lithium-containing mouthwash — The main ingredients of lithium-containing mouthwash are lithium carbonate and citric acid. A total of 5 concentration gradients of lithium-containing mouthwash are set, including 0.03, 0.06, 0.10, 0.15 and 0.30 mol/L. Mouthwash is used to gargle and left in the mouth for 5 min to be spat out three times a day from the first day of radiotherapy up to the end of treatment.
  Arms: 0.30 mol/L lithium mouthwash
Drug: Plcacebo mouthwash — Placebo Mouthwash is mainly composed of citric acid and sodium hydroxide, transparent colorless liquid. Mouthwash is used to gargle and left in the mouth for 5 min to be spat out three times a day from the first day of radiotherapy up to the end of treatment.
  Arms: Placebo mouthwash
Drug: lithium-containing mouthwash — Effective lithium salt concentrations screened in the Phase I trial is used as active interventions in this group of interventions. Mouthwash is used to gargle and left in the mouth for 5 min to be spat out three times a day from the first day of radiotherapy up to the end of treatment.
  Arms: Lithium mouthwash

SUMMARY:
To evaluate the efficacy and safety of lithium-containing mouthwash for prevention and treatment of oral mucositis and dysgeusia in patients undergoing radiotherapy for malignant head and neck tumors.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the efficacy and safety of lithium-containing mouthwash in reducing the incidence, duration, and severity of severe oral mucositis (SOM) , and the incidence of dysgeusia. The main questions it aims to answer are whether lithium-containing mouthwash can effectively prevent and treat radiation-induced oral mucositis and dysgeusia, and whether it will cause adverse events in patients undergoing radiotherapy.

Participants will be instructed to use lithium-containing mouthwash or placebo mouthwash three times daily from the beginning to the end of RT.

Researchers will compare lithium-containing mouthwash group and placebo group to see if lithium-containing mouthwash are beneficial in preventing and treating oral mucositis and dysgeusia in patients undergoing radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

Patients pathologically diagnosed with non-metastatic head and neck malignant tumors; Aged 18-80 years; Eastern Cooperative Oncology Group performance status of ≤2; Planning to receive definitive RT or postoperative adjuvant RT; Normal liver, kidney and bone marrow function; Sign informed consent.

Exclusion Criteria:

Known to be allergic to lithium or other components of mouthwash or severe allergic constitution; Poor oral hygiene and/or severe periodontal diseases; Any previous RT to the head and neck region, Severe kidney disease, severe cardiovascular disease, myasthenia gravis, Parkinson's disease or epilepsy; Recent use or current use of diuretics or other drugs known to interact with lithium; Deemed unsuitable for the study by the investigators (concomitant with any other severe diseases).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
The incidence of Severe Oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy
  Oral mucositis is assessed by trained physicians according to World Health Organization (WHO) oral toxicity Scale.

SECONDARY OUTCOMES:
Xerostomia | 1 week before radiotherapy ; at the middle of radiotherapy (3 weeks after the start of radiotherapy) ; at the end of radiotherapy (the last radiation dose received, usually 6 or 6.5 weeks); and 1, 3, 6, 9 and 12 months after the end of radiotherapy
  Patients self-rated xerostomia according to summated xerostomia inventory (SXI), and researchers measured saliva flow rates.
Patients' quality of life assessment of EORTC QLQ-C30 and H&N35 questionnaires. | 1 week before radiotherapy; at the end of radiotherapy(the last radiation dose received, usually 6 or 6.5 weeks); ; and 1, 3, 6, 9 and 12 months after the end of radiotherapy
  EORTC QLQ-C30 and H&N35 questionnaires
Adverse events | From the first day of radiotherapy to the day of the last radiation dose received, usually 6 or 6.5 weeks
  Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version
Mouth and throat soreness (MTS) scores | The time period is the period from the start of radiotherapy to the completion of radiotherapy.The evaluation period is approximately 6 weeks and 6 1/2 weeks
  Patients report mouth and throat soreness (MTS) scores (Likert scale 1 to 5) via the oral mucositis weekly questionnaire （OMWQ）. Higher score indicates more severe symptoms.
The duration of Severe Oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy
  The first determination of SOM to the first instance of non-severe OM (WHO grade <3), without a subsequent instance of SOM. Patients without observed SOM were assigned a duration of 0 days.
The time to onset of Severe Oral mucositis (WHO grade ≥3) | From the start of radiotherapy to 8 weeks after completion of radiotherapy
  Time from the first day of radiotherapy to the first determination of SOM. Patients without observed SOM were assigned onset days of 6 or 6.5 weeks.
Taste function | 1 week before radiotherapy ; at the middle of radiotherapy (3 weeks after the start of radiotherapy) ; at the end of radiotherapy (the last radiation dose received, usually 6 or 6.5 weeks); and 1, 3, 6, 9 and 12 months after the end of radiotherapy
  Patients self-rated dysgeusia, Electrogustometer test and taste strips test.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No